CLINICAL TRIAL: NCT06545331
Title: A Dose-Escalation and Expansion Study of XB010 as a Single Agent and Combination Therapy in Subjects With Locally Advanced or Metastatic Solid Tumors
Brief Title: Study of XB010 in Subjects With Solid Tumors
Acronym: DELTA-101
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XB010-101
Record Dates: First submitted 2024-07-29; First posted 2024-08-09 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Locally Advanced or Metastatic Solid Tumors; Esophageal Squamous Cell Cancer; Head and Neck Squamous Cell Cancer; NSCLC (Non-small Cell Lung Cancer); Hormone-receptor-positive Breast Cancer; Triple Negative Breast Cancer (TNBC)
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Carcinoma, Non-Small-Cell Lung; Triple Negative Breast Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- XB010 Single-Agent Dose Escalation Cohorts (Experimental): XB010 will be administered at escalating dose levels every 3 weeks in cohorts of 3-12 subjects
  Interventions: Drug: XB010
- XB010 + Pembrolizumab Dose Escalation Cohorts (Experimental): XB010+Pembrolizumab will be administered at escalating dose levels every 3 weeks in cohorts of 3-12 subjects
  Interventions: Drug: XB010; Drug: Pembrolizumab
- XB010 Single-Agent Dose Expansion Cohorts (Experimental): XB010 will be administered at the recommended dose for expansion (RDE) every 3 weeks in the following tumor-specific cohorts: non-small cell lung cancer (NSCLC), hormone-receptor-positive breast cancer (HR+BC), head and neck squamous cell cancer (HNSCC), esophageal squamous cell cancer (ESCC), endometrial cancer (EC) and triple-negative breast cancer (TNBC)
  Interventions: Drug: XB010

INTERVENTIONS:
Drug: XB010 — IV administration of XB010
Drug: Pembrolizumab — IV administration of Pembrolizumab
  Arms: XB010 + Pembrolizumab Dose Escalation Cohorts

SUMMARY:
This is a FIH study is to evaluate the safety, tolerability, PK, immunogenicity, and preliminary antitumor activity of XB010 as a single agent and in combination with pembrolizumab in subjects with locally advanced or metastatic solid tumors for whom alternative therapies do not exist or available therapies are intolerable or no longer effective.

DETAILED DESCRIPTION:
This study consists of Dose-Escalation and Cohort-Expansion Stages. The Dose-Escalation Stage is designed to determine the maximum tolerated dose (MTD) and/or recommended dosage(s) for expansion (RDE[s]) of XB010 as a single agent, and to evaluate XB010 monotherapy RDE(s) in combination with pembrolizumab. The Cohort-Expansion Stage is designed to explore the clinical activity and further characterize the safety and tolerability of XB010 as monotherapy in multiple tumor-specific cohorts.

ELIGIBILITY:
* Age 18 years or older on the day of consent.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1.
* Adequate organ and marrow function.
* Cytologically or histologically and radiologically confirmed solid tumor that is inoperable, locally advanced, metastatic, or recurrent.

  * The Cohort Expansion stage will enroll subjects with multiple tumor types (non-small cell lung cancer, hormone-receptor-positive breast cancer, head and neck cancer, esophageal squamous cell, triple-negative breast cancer).
* Capable of understanding and complying with the protocol requirements and must have signed the informed consent document.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Estimated)
Dates: Start 2024-08-06 (Actual); Primary Completion 2026-11-23 (Estimated); Study Completion 2027-10-20 (Estimated)

PRIMARY OUTCOMES:
Dose-Escalation Stage: Maximum tolerated dose (MTD) and/or Recommended dose(s) for Expansion [RDE(s)] for XB010 | 18 months
  To determine the MTD and/or RDE(s) for further evaluation of IV administration of XB010 alone and in combination therapy.
Dose-Escalation Stage: Safety of XB010 | 18 months
  To evaluate the safety of XB010 alone and in combination therapy through the evaluation of incidence and severity of nonserious adverse events (AEs) and serious adverse events (SAEs)
Dose-Escalation Stage: Duration of exposure of XB010 [Tolerability] | 18 months
  To evaluate the tolerability of XB010 alone and in combination therapy through the evaluation of the duration of exposure of each component
Dose-Escalation Stage: Dose intensity of XB010 [Tolerability] | 18 months
  To evaluate the tolerability of XB010 alone and in combination therapy through the evaluation of the dose intensity of each component
Cohort-Expansion Stage: Preliminary antitumor activity of XB010 | 24 months
  Objective Response Rate (ORR) as assessed by the Investigator per RECIST 1.1

SECONDARY OUTCOMES:
Dose-Escalation Stage: Maximum Plasma Concentration (Cmax) of XB010 | 18 Months
  To evaluate the maximum plasma concentration of XB010 alone and in combination.
Dose-Escalation Stage: Time to Maximum Plasma Concentration (Tmax) of XB010 | 18 Months
  To evaluate the time to maximum plasma concentration of XB010 alone and in combination.
Dose-Escalation Stage: Clearance of XB010 | 18 Months
  To evaluate the volume of plasma cleared of XB010 alone and in combination for a specified time period
Dose-Escalation Stage: Area Under the Plasma Concentration Curve (AUC) of XB010 | 18 Months
  To measure the Area Under the Plasma Concentration Curve of XB010 alone and in combination
Dose-Escalation Stage: Minimum Plasma Concentration (Cmin) of XB010 | 18 Months
  To evaluate the minimum plasma concentration of XB010 alone and in combination
Dose-Escalation Stage: Immunogenicity of XB010 | 18 Months
  To assess the immunogenicity of XB010 alone and in combination as measured by anti-drug antibody (ADA) analysis
Cohort-Expansion Stage: Duration of exposure of XB010 [Tolerability] | 24 Months
  To evaluate the tolerability of XB010 through the evaluation of the duration of exposure
Cohort-Expansion Stage: Dose intensity of XB010 [Tolerability] | 24 Months
  To evaluate the tolerability of XB010 through the evaluation of the dose intensity
Cohort-Expansion Stage: Maximum Plasma Concentration (Cmax) of XB010 | 24 Months
  To evaluate the maximum plasma concentration of XB010
Cohort-Expansion Stage: Time to Maximum Plasma Concentration (Tmax) of XB010 | 24 Months
  To evaluate the time to maximum plasma concentration of XB010
Cohort-Expansion Stage: Clearance of XB010 | 24 Months
  To evaluate the volume of plasma cleared of XB010 for a specified time period
Cohort-Expansion Stage: Area Under the Plasma Concentration Curve (AUC) of XB010 | 24 Months
  To measure the Area Under the Plasma Concentration Curve of XB010
Cohort-Expansion Stage: Minimum Plasma Concentration (Cmin) of XB010 | 24 Months
  To evaluate the minimum plasma concentration of XB010
Cohort-Expansion Stage: Immunogenicity of XB010 | 24 Months
  To assess the immunogenicity of XB010 as measured by anti-drug antibody (ADA) analysis

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Exelixis
Locations (15):
- United States (13):
  - Exelixis Clinical Site #4, Irvine, California
  - Exelixis Clinical Site #10, Washington D.C., District of Columbia
  - Exelixis Clinical Site #12, Atlanta, Georgia
  - Exelixis Clinical Site #15, Chicago, Illinois
  - Exelixis Clinical Site #5, St Louis, Missouri
  - Exelixis Clinical Site #3, Huntersville, North Carolina
  - Exelixis Clinical Site #6, Oklahoma City, Oklahoma
  - Exelixis Clinical Site #9, Nashville, Tennessee
  - Exelixis Clinical Site #1, Austin, Texas
  - Exelixis Clinical Site #7, Dallas, Texas
  - Exelixis Clinical Site #8, Houston, Texas
  - Exelixis Clinical Site #11, Fairfax, Virginia
  - Exelixis Clinical Site #2, Fairfax, Virginia
- United Kingdom (2):
  - Exelixis Clinical Site #13, London, England
  - Exelixis Clinical Site #14, Manchester, England

IPD SHARING:
Plan to Share IPD: No